CLINICAL TRIAL: NCT05988957
Title: Perspectives on Using a Nutrition-focused Approach When Initiating Continuous Glucose Monitoring in People With Type 2 Diabetes: a Qualitative Study
Brief Title: Nutrition-Focused Approach During CGM Initiation: A Qualitative Study
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Holly Willis, PhD, RDN, CDCES, HealthPartners Institute
Other Study IDs: A22-279
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: continuous glucose monitor; CGM; nutrition; qualitative interview
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-structured interviews using an IRB-approved interview guide — A single, semi-structured interview will be conducted using an IRB-approved interview guide. The interviews will be approximately 30 minutes total.

SUMMARY:
The purpose of the qualitative research is to provide a deeper understanding of the perspectives of people with type 2 diabetes (T2D) who received a nutrition-focused approach (NFA) when initiating continuous glucose monitor (CGM).

DETAILED DESCRIPTION:
The purpose of the qualitative research is to provide a deeper understanding of the perspectives of people with T2D who received the NFA when initiating CGM.

A single 30-minute semi-structured interview will be conducted in approximately 15 people who have completed participation in the A21-292 study (also called the My Diabetes Study).

The My Diabetes Study, is a randomized clinical trial to assess the impact of using a NFA or a self-directed approach during CGM initiation. The NFA was developed specifically for the randomized clinical trial study.

ELIGIBILITY:
Inclusion Criteria:

* Participant was randomized to the nutrition-focused approach arm of the My Diabetes study
* Participant completed all required study visits in the My Diabetes study; this includes the baseline visit, the two intervention visits, and the study completion visit
* Participant had at least 70% "Time CGM Active" on a 10-day Dexcom Clarity Report at study completion visit
* Participant is willing to be recorded during the interview

Exclusion Criteria:

* Participant was randomized to the self-directed approach study arm of the My Diabetes study
* Participant is deemed unsuitable for participation due to any cause as determined by the Investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults who have met inclusion criteria for the My Diabetes study and who have completed the nutrition-focused approach arm of the study may be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Willis, PhD, Principal Investigator — HealthPartners Institute; International Diabetes Center
Locations (1):
- HealthPartners Institute dba International Diabetes Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Interviews were completed between September 2023 and March 2024.
Pre-assignment Details: All participants had to meet inclusion criteria for the larger UNITE study (NCT05928572), be randomly assigned to the nutrition-focused approach arm, complete all components of the 2-month UNITE study intervention, have adequate CGM data at the final postintervention assessment, and be willing to participate in a recorded interview.
Groups:
- Semi-structured Inteviewees: People who participated in the semi-structured interviews
Period: Overall Study
Arm/Group | Semi-structured Inteviewees
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Information about all of 15 people who participated in the interviews are provided.
Groups:
- Semi-structured Inteviews: People who participated in the semi-structured interviews
Arm/Group | Semi-structured Inteviews
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — age in years was collected by assessing participants birthday at the time of the interview
  years | 64.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants were asked to self-identify thier sex and this information was recorded on source documents
  Participants
    Female | 6
    Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Glycated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent of glycated hemoglobin] — HbA1c was assessed during the parent UNITE study; this was done by collecting a small blood sample via a venous draw. The value was taken from the electronic medical record.
  percent of glycated hemoglobin | 7.5 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Describe CGM Data Use by 15 of the Participants During the UNITE/MyDiabetes Study
Description: 30 minute interviews with each participant were transcribed and thematic coding was used to describe how participants in the My Diabetes Study used their CGM data when making food-related decisions after receiving a nutrition-focused approach during CGM initiation. Narrative summaries of the data were written up to describe the findings from all 15 participants. No objective outcome data is available to present in the outcome measure data table.
Time Frame: Immediately following the 2-month study completion visit in the My Diabetes study.
Population: People who met inclusion/exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Semi-structured Inteviewees
Number analyzed (Participants) | 15
Participants
  Number of people completing interview | 15
  Number of participants who used CGM to make food-related decisions | 15

2. Secondary Outcome: Describe the Overall Experience of 15 Participants Receiving a Nutrition-focused Approach During CGM Initiation During the UNITE/MyDiabetes Study
Description: 30 minute interviews with each participant were transcribed and thematic coding was used to describe how participants with T2D in the My Diabetes Study experienced the use of a nutrition-focused approach and its associated nutrition-focused CGM initiation materials during CGM initiation. Narrative summaries of the data were written up to describe the findings from all 15 participants. No objective outcome data is available to present in the outcome measure data table.
Time Frame: Immediately following the 2-month study completion visit in the My Diabetes study.
Population: People who met inclusion/exclusion criteria were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Semi-structured Inteviewees
Number analyzed (Participants) | 15
Participants
  Number of Participants | 15
  Number who agreed pairing nutrition information with CGM initiation was helpful for diabetes care | 15

ADVERSE EVENTS:
Time Frame: This was a qualitative interview at one point in time. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: This was a qualitative interview. No adverse events were expected.
Arm/Group | Semi-structured Inteviewees
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
One limitation is that this research did not assess the perspectives and behaviors of people with T2D who initiated CGM without an Nutrition focused approach (eg, with a self-directed approach). Thus, it is unclear whether people without a Nutrition focused approach during CGM initiation would have similar experiences and report similar views during CGM initiation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT05988957/Prot_000.pdf